CLINICAL TRIAL: NCT03809494
Title: Clinical Study of the Use of an Autologous Blood Filtration Device in the Treatment of Critical Limb Ischemia
Brief Title: HemaTrate™ in the Treatment of Critical Limb Ischemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has stopped early due to enrollment challenges related largely to the current pandemic
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-03
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Critical Limb Ischemia; Ischemia
Keywords: lower extremity; Peripheral Arterial Disease; Ischemia; Peripheral Blood Stem Cell Transplantation; Leukocytes, Mononuclear; Transplantation, Autologous
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Ischemia; Peripheral Arterial Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The investigator for this study is the person that will be performing the injections throughout the study and will know the participant's treatment (TNC or saline). The investigator that is aware of the participant's treatment will not be performing the follow-up visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Patients assigned to the treatment arm will be injected with autologous concentrated total nucleated cells (TNCs) three times at six week intervals.
  Interventions: Device: HemaTrate™ Blood Filtration system
- Saline (Control Arm) (Placebo Comparator): Patients assigned to the control arm will be injected with saline three times at six week intervals.
  Interventions: Other: Saline

INTERVENTIONS:
Device: HemaTrate™ Blood Filtration system — Anticoagulated whole blood is loaded into the filtration system. During gravity filtration, the majority of platelets, plasma, and red blood cells pass through the filter into a filtrate bag. The TNCs are captured in the filter material and recovered via a back-flush with 0.9 % saline into a syringe.
  Arms: Treatment Arm
Other: Saline — Normal (0.9%) saline
  Arms: Saline (Control Arm)

SUMMARY:
The primary objective of this study is to evaluate the performance of the HemaTrate™ Blood Filtration system in the treatment of critical limb ischemia. The primary endpoint measure is comparing the percentage of patients between the treatment arm and control arm who have freedom from major amputation, arterial intervention below the knee, and death through 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Critical Limb Ischemia in the study leg with ischemic rest pain and/or ulcer/minor tissue loss (Rutherford 4 or 5)
2. Previously failed an endovascular or surgical treatment of the study lower leg and is not being considered for additional intervention within the next 3 months OR is unsuitable for revascularization

Exclusion Criteria:

1. Simultaneously participating in another investigational study (e.g., drug or device)
2. Pregnant or breastfeeding, or planning to become pregnant within the next 12 months
3. Major surgery (open cardiac, vascular, or abdominal procedure) within the past 90 days
4. Endovascular intervention within the past 30 days
5. Current dialysis, or expected to need dialysis within the next 12 months
6. Previous above the ankle amputation in the study leg

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Freedom from vascular or endovascular arterial intervention below the knee of the study leg | 12 months
  Percent of patients that have vascular or endovascular arterial intervention reported below the knee of the study leg
Freedom from major amputation of the study leg | 12 months
  Percent of patients that have any amputation above the ankle of the study leg
Death | 12 months
  Percent of patients that exit due to death

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Modarai, PhD, FRCS, Study Chair — St Thomas' Hospital; Václav Procházka, MD, PhD, MSc, Study Chair — University Hospital Ostrava; Giulio Pompilio, MD, PhD, Study Chair — Centro Cardiologico Monzino IRCCS
Locations (3):
- United Kingdom (3):
  - Manchester Royal Infirmary, Manchester Vascular Centre, Manchester, Great Britian
  - The Leeds Teaching Hospital NHS Trust, Leeds, West Yorkshire
  - St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after publication of the results from this study and ending 5 years after initial publication. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.